CLINICAL TRIAL: NCT05878756
Title: Effects of Additional Functional Strength Training on Mobility in Children With Hemiplegic Cerebral Palsy,A Randomized Control Trail
Brief Title: Effects of Additional Functional Strength Training on Mobility in Children With Hemiplegic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Health Education Research Foundation (HERF) (Other)
Responsible Party: Principal Investigator, Mamoona Tasleem Afzal, Mamoona Tasleem Afzal, Health Education Research Foundation (HERF)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YIRS/1666
Record Dates: First submitted 2023-05-19; First posted 2023-05-26 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Hemiplegic Cerebral Palsy; Mobility
Keywords: Cerebral palsy; Functional strength training; Mobility; GMFC; GMFM
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional strength training (Experimental): With conventional therapy,the ten tasks were STS, one leg standing, weight shifting(from one side of body to other), step-ups, lateral step-ups, squatting against wall, picking an object from standing position, walking forward, walking backward and kicking the ball preform from the patient 5 days per week for 4 weeks.
  Interventions: Other: Functional Strength Training
- Conventional therapy (Active Comparator): passive and active range of motion exercises,Stretching and strengthening exercise 5 days per week for 4 weeks.
  Interventions: Other: Functional Strength Training

INTERVENTIONS:
Other: Functional Strength Training — In addition to conventional therapy, experimental group was also given functional strength training program. Functional strength training was given as home program consisting of ten tasks.The ten tasks were STS, one leg standing, weight shifting(from one side of body to other), step-ups, lateral step-ups, squatting against wall, picking an object from standing position, walking forward, walking backward and kicking the ball.
  Other Names: conventional therapy

SUMMARY:
The randomized control trail was to determine the effects of additional functional Strength Training on mobility in Children with Hemiplegic Cerebral Palsy.

DETAILED DESCRIPTION:
The aim of functional physiotherapy is to train the child by emphasizing him to learn motor abilities. These motor abilities are those that are thought to be though either by children with cerebral palsy or their parents. Functional activities are learned by the repetitive practice of goal-oriented tasks in a given functional situation. This approach instead of focusing on normality, it focuses on functionality. In this way, it is very necessary for the child to practice a given task functionally rather than normally.No studies have been done to improve mobility and strength in lower limb in children with hemiplegia cerebral palsy. So for this reason, this study is conducted to investigate the effects of additional functional Strength Training on mobility in Children with Hemiplegic Cerebral Palsy.In this way we can make these children an active participant of the society.

ELIGIBILITY:
Inclusion Criteria:

children who didnot use the assistive device children who follow the commands children who did not treated in any other rehabilitation center

Exclusion Criteria:

children with any other diagnosis other than CP children with fixed contractures children underwent surgery children who received Botulinum Toxin

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Gross Motor Function Measure (GMFM) | Data was collected at Baseline and after 4 weeks
  GMFM is used to evaluate change that occurs over time in the gross motor function of children with cerebral palsy.
Gross Motor Function Classification System (GMFCS) | Data was collected at Baseline and after 4 weeks
  The GMFCS, or Gross Motor Function Classification System, is a five-level classification that differentiates children with cerebral palsy based on the child's current gross motor abilities, limitations in gross motor function, and need for assistive technology and wheeled mobility.

SECONDARY OUTCOMES:
Five time sit to stand (FTSST). | Data was collected at Baseline and after 4 weeks
  Used to asses functional lower extremity strength, transitional movements, balance, and fall risk

CONTACTS AND LOCATIONS:
Locations (1):
- Yusra Institute of Rehablitation Science, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No